CLINICAL TRIAL: NCT02716636
Title: Fast Versus Slow Tenaculum Placement for Office Procedures: A Randomized Controlled Trial
Brief Title: Fast Versus Slow Tenaculum Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbey Hardy-Fairbanks (Other)
Responsible Party: Sponsor-Investigator, Abbey Hardy-Fairbanks, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201509756
Record Dates: First submitted 2015-11-17; First posted 2016-03-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: IUD Insertion Complication; Endometrial Diseases
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast placement (No Intervention): Placement of the tenaculum quickly and without avoiding ratchet
- Slow placement of the tenaculum (Experimental): Placement of the tenaculum over a 7-10 second time frame and not allowing the tenaculum to ratchet audibly.
  Interventions: Procedure: Slow placement of the tenaculum

INTERVENTIONS:
Procedure: Slow placement of the tenaculum — Slow placement of the tenaculum on the cervix
  Arms: Slow placement of the tenaculum

SUMMARY:
The purpose of the study is to investigate whether the speed of tenaculum placement affects perceived patient pain during office transcervical procedures.

DETAILED DESCRIPTION:
IUD insertion and endometrial biopsies are commonly performed in office procedures that use a tenaculum to stabilize the cervix. Patient's often complain that tenaculum placement is one of the most uncomfortable parts of these procedures. Patient's who agree to be in the study will be randomized into one of two groups, either slow tenaculum placement or fast tenaculum placement. Throughout the procedure patient's will be asked to rate the amount of pain they are experiencing using a visual analog scale. The researchers will then compare the two groups. The providers will also rate what they perceived the patient's pain to be with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Clinic provider plans a transcervical procedure (IUD placement or endometrial biopsy)
* English speaking and able to consent

Exclusion Criteria:

* Incarcerated
* Prior LEEP (loop electrosurgical excision procedure), cryo (cryotherapy) or CKC (cold knife cone) of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Pain with tenaculum placement assessed using a VAS scale | procedure
  Subjects will record their pain on a paper VAS scale at the time of the procedure only. This is the only data collection point for this measure.

SECONDARY OUTCOMES:
Overall pain perception assessed using a VAS scale | procedure
  Subjects will record their pain on a paper VAS scale at the time of the procedure only. This is the only data collection point for this measure.
Provider perception of patient pain assessed using a VAS scale | procedure
  Providers will record their pain on a paper VAS scale at the time of the procedure only. This is the only data collection point for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey J Hardy-Fairbanks, MD, Principal Investigator — University of Iowa